CLINICAL TRIAL: NCT06479785
Title: Effects of an Educational Intervention Program on Lung Function and Ergonomic Hazards Among Marble Factory Workers: Quasi-experimental Study
Brief Title: Effects of an Educational Intervention Program on Marble Factory Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Waseem Ullah
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Diseases
Keywords: lung function, ergonomic hazards, marble factory workers
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention program on machine workers (Experimental): Use proper protective gears like mask, glasses, glove and proper foot wear. Maintain proper posture. Avoid repetitive movement.
  Interventions: Other: Educational Intervention Program for machine workers
- Educational intervention program on manual workers (Experimental): Use proper protective gears like mask, glasses, glove and proper foot wear. Maintain proper posture during heavy load lifting. Take breaks during prolong period of work.
  Interventions: Other: Educational Intervention Program for manual workers

INTERVENTIONS:
Other: Educational Intervention Program for machine workers — A detailed Educational Intervention Program for marble factory workers working on Machines.
  Arms: Educational intervention program on machine workers
Other: Educational Intervention Program for manual workers — A detailed Educational Intervention Program for marble factory workers working manually.
  Arms: Educational intervention program on manual workers

SUMMARY:
Marble cutting exposes workers to dust, increasing risk of lung diseases like asthma, COPD, silicosis, and asbestosis. Many marble cutters in rural areas lack awareness of these risks and work without proper protection. Khyber Pakhtunkhwa has over 4000 marble factories employing over a million laborers, mostly unskilled and vulnerable. Workers face health risks from heavy lifting, poor posture, and respirable dust. Ergonomic disorders are also common due to poorly designed workstations, repetitive motions, and straining postures. Musculoskeletal Symptoms (MSS) can progress into Musculoskeletal Disorders (MSDs), affecting worker well-being and productivity. Findings can inform targeted educational programs and interventions to improve respiratory health and reduce ergonomic risks in the marble industry.

DETAILED DESCRIPTION:
Occupational hazards, such as dust exposure during marble cutting, can significantly increase the risk of lung diseases in workers. This includes common ailments such as asthma and Chronic Obstructive Pulmonary Disease (COPD), as well as more serious conditions such as silicosis and asbestosis. Unfortunately, many marble cutters from rural areas may not be aware of these health risks, which can lead to them working without proper protection. Heavy load lifting, poor work posture, and the production of respirable dust in marble factories contribute to the health risks faced by these workers. Just like dust exposure during marble cutting can harm a worker's lungs, similarly, working in this industry carries a high risk of ergonomic disorders. According to the Bureau of Labor Statistics, ergonomic risk factors are responsible for 35% of workplace injuries in 2021, resulting in MSDs. An extensive amount of research has been conducted globally; however, limited literature exists on this particular topic in Khyber Pakhtunkhwa, specifically in Peshawar. The findings of the study can help inform the development and implementation of targeted educational programs and interventions aimed at improving respiratory health and reducing ergonomic risks in the marble industry.

ELIGIBILITY:
Inclusion Criteria:

* Adult male marble factory workers,
* Age 20-55years
* Working for more than 1year
* Working time(hours): minimum 06 hours daily

Exclusion Criteria:

* Workers with pre-existing lung diseases
* Workers with any other occupational hazard
* Workers who are not willing to participate in the study

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | 4 weeks
  Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced vital capacity (FVC) | 4 weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
Forced expiratory volume in 1sec (FEV1) | 4 weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal

SECONDARY OUTCOMES:
Rapid Upper Limb Assessment (RULA) | 4 Weeks
  RULA evaluates the exposure to posture and force/external load as well as repeated and static posture effects.
Rapid Entire Body Assessment (REBA) | 4 Weeks
  REBA evaluates the exposure to posture and force/external load as well as repeated and static posture effects. The REBA has two additional assessment factors of coupling and dynamic loading effects, compared to the RULA

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Marble factories in Peshawar, Islamabad, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butt IM, Mustafa T, Rauf S, Razzaq A, Anwer J. Pulmonary function parameters among marble industry workers in Lahore, Pakistan. F1000Res. 2021 Sep 17;10:938. doi: 10.12688/f1000research.52749.1. eCollection 2021. PMID 34868564
- [Background] Chen CH, Tsai PJ, Chang WW, Chen CY, Chen CY, Yates D, Guo YL. Dose-response relationship between lung function and chest imaging response to silica exposures in artificial stone manufacturing workers. Environ Health. 2024 Mar 2;23(1):25. doi: 10.1186/s12940-024-01067-1. PMID 38429786